CLINICAL TRIAL: NCT01932879
Title: Blackberry Polyphenol Intake and Fuel Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Janet Novotny, Research Physiologist, USDA Beltsville Human Nutrition Research Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: HS44
Record Dates: First submitted 2013-08-27; First posted 2013-08-30 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Fuel Management
MeSH Terms: interventions — Gels

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Blackberry (Experimental): Participants will consume blackberries twice/day as part of a 1-week controlled diet.
  Interventions: Other: Blackberry
- Control (Other): Participants will consume jello twice/day as part of a 1-week controlled diet.
  Interventions: Other: Jello

INTERVENTIONS:
Other: Blackberry — Participants will be fed a higher fat, typical American diet for two 1-week periods. Participants must consume only and all food provided during the intervention periods.
  Arms: Blackberry
Other: Jello
  Arms: Control

SUMMARY:
Studies in animals have suggested that berry preparations or anthocyanin-rich berry extracts can reduce body fatness. Previous studies with tea catechins, which belong to the flavonoid class of chemicals as do anthocyanins, suggest that these compounds can alter fat oxidation, and this may be the mechanism by which body fatness is influenced by anthocyanin intake. Well-controlled studies in humans are lacking.

ELIGIBILITY:
Exclusion Criteria:

* Younger than 25 years old or older than 75 years old
* Female
* Use of blood-thinning medications such as Coumadin (warfarin), Dicumarol (dicumarol), or Miradon (anisinidione)
* Presence of any gastrointestinal disease, metabolic disease, or malabsorption syndromes that may interfere with the study goals
* Have been pregnant during the previous 12 months, are currently pregnant or lactating, or plan to become pregnant during the study
* Type 2 diabetes requiring the use of oral antidiabetic agents or insulin
* Fasting triglycerides greater than 300 mg/dL
* Fasting glucose greater than 126 mg/dL
* History of eating disorders or other dietary patterns which are not consistent with the dietary intervention (e.g., vegetarians, very low fat diets, high protein diets)
* Use of prescription or over-the-counter antiobesity medications or supplements (e.g., phenylpropanalamine, ephedrine, caffeine) during and for at least 6 months prior to the start of the study or a history of a surgical intervention for obesity
* Active cardiovascular disease (such as a heart attack or procedure within the past three months or participation in a cardiac rehabilitation program within the last three months, stroke, or history/treatment for transient ischemic attacks in the past three months, or documented history of pulmonary embolus in the past six months).
* Use of any tobacco products in past 3 months
* Use of oral or IV antibiotics during the month preceding the study
* Unwillingness to abstain from herbal supplements for two weeks prior to the study and during the study
* Known (self-reported) allergy or adverse reaction to blackberries
* Unable or unwilling to give informed consent or communicate with study staff
* Self-report of alcohol or substance abuse within the past twelve months and/or current acute treatment or rehabilitation program for these problems (Long-term participation in Alcoholics Anonymous is not an exclusion)
* Other medical, psychiatric, or behavioral factors that in the judgment of the Principal Investigator may interfere with study participation or the ability to follow the intervention protocol

Ages: 25 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-07; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Substrate oxidation | 23.5 hours
  Participants will stay in a room calorimeter for 23.5 hours.

SECONDARY OUTCOMES:
Glucose tolerance test | -15, 0, 30, 60, 90, 120, 180, 240 minutes
  Blood will be collected at the end of each diet period, at the following times before and after breakfast: -15, 0, 30, 60, 90, 120, 180, 240 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- USDA Beltsville Human Nutrition Research Center, Beltsville, Maryland, United States